CLINICAL TRIAL: NCT06908980
Title: CHOLE-POSSUM PRO Validation for Prediction of Mortality After Cholecystectomy for Acute Calculous Cholecystitis: Protocol for a Prospective Multicenter Observational Study
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Luca Ansaloni, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: CHOLE-POSSUM PRO
Record Dates: First submitted 2025-03-22; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Acute Calculous Cholecystitis Candidate to Early Cholecystectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients who receive a diagnosis of ACC as defined by TG18 criteria and with ACC

SUMMARY:
CHOLE-POSSUM PRO is a prospective multicenter observational study on patients with ACC candidate to EC. The rationale of the study is to validate the CHOLE-POSSUM PRO SCORE for 30-day mortality in this population.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of ACC as defined by TG18 criteria
* be ACC candidate to EC during the index admission* (* All the patients treated with initial open cholecystectomy, those who undergo ELC, those with conversion from laparoscopic to open cholecystectomy or those who undergo bail out procedures (e.g. subtotal cholecystectomy) will be included.)
* be ≥ 18 years old
* be stratified for the risk of CBDS according to the Israelian Score (29), and, in case of confirmation of CBDS receive pre-operative ERCP
* provide signed and dated informed consent form
* willing to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* pregnancy or lactation
* acute cholecystitis not related to a gallstone etiology
* onset of symptoms >10 days before cholecystectomy** (** Patients with ACC associated with common bile duct stones who underwent pre-operative ERCP could be included if they receive EC within 10 days from onset of symptoms)
* concomitant pancreatitis
* intraoperative treatment of common bile duct stones
* anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive a diagnosis of ACC as defined by TG18 criteria and with ACC candidate to EC during the index admission
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-10-11 (Estimated); Study Completion 2025-10-11 (Estimated)

PRIMARY OUTCOMES:
The AUC-ROC for 30-days mortality computed in the validating cohort | Day 30

SECONDARY OUTCOMES:
The AUC-ROC for 30-days major complications (Clavien-Dindo ≥3) rate computed in the validating cohort | Day 30

OTHER OUTCOMES:
Intraoperative complications rate | through study completion, an average of 2 years
Duration of surgery | immediately after the surgery
Conversion rate | through study completion, an average of 2 years
Length of stay (LOS) | through study completion, an average of 2 years
30-days readmission rate | Day 30
Result of blood and bile cultures | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Italy